CLINICAL TRIAL: NCT01707563
Title: Correlations' Study Between Variability of Expression in FBN1 Gene and Clinical Features in Marfan Patients.
Brief Title: Clinical Variability in Marfan Syndrome
Acronym: Variarfan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hospices Civils de Lyon (Other); Banque de cellules cochin (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: P071009
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2010-12

CONDITIONS: Marfan Syndrome
Keywords: Marfan syndrome; Variability; Fibrillin 1; clinical expression
MeSH Terms: conditions — Marfan Syndrome; Arachnodactyly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marfan patients (Other): Study participants were recruited between 11/2009 and 10/2011, among adult patients consulting in the Multidisciplinary Marfan Clinic of our University Hospital, and having a known mutation in the FBN1 gene. There, patients are evaluated by geneticists, rheumatologists, cardiologists, and ophthalmologists. Systematic slit-lamp examination, cardiac ultrasonography, and radiological investigations are also performed. A skin punch biopsy was used to establish a fibroblast cell culture. We determined mRNA levels for FBN1 and compared it to the clinical involvement.
  Interventions: Procedure: skin punch biopsy and molecular biology
- control patients (Other): Fibroblasts were obtained from non Marfan patients (cell bank). We determineed mRNA level for FBN1 for each allele.
  Interventions: Other: fibroblast culture and molecular biology

INTERVENTIONS:
Procedure: skin punch biopsy and molecular biology
  Arms: Marfan patients
Other: fibroblast culture and molecular biology
  Arms: control patients

SUMMARY:
Marfan syndrome is an autosomal dominant connective tissue disorder caused by mutations in the fibrillin-1 gene (FBN1). Penetrance of FBN1 mutations is complete but intra and inter familial clinical expressivity is extremely variable. The underlying mechanisms for variability are not understood. An interesting mechanism is that the expression level of the wild type and/or mutated allele may play a role in the determination of variability.

Principal objective: To evaluate in Marfan patients, if FBN1 expression level (non-mutated or mutated allele) modulates the clinical expression of the disease.

Judgment criteria : Correlation allelic expression level-phenotype Perspectives : To search the predictive factors of severity in order to ameliorate precocity of taking care.

DETAILED DESCRIPTION:
Marfan syndrome is an autosomal dominant connective tissue disorder caused by mutations in the fibrillin-1 gene (FBN1). Penetrance of FBN1 mutations is complete but intra and inter familial clinical expressivity is extremely variable. The underlying mechanisms for variability are not understood. An interesting mechanism is that the expression level of the wild type and/or mutated allele may play a role in the determination of variability.

Principal objective : To evaluate in Marfan patients, if FBN1 expression level (non-mutated or mutated allele) modulates the clinical expression of the disease in individuals from families with clinical variability (intrafamilial) and in independant probands (interfamilial).

Judgment criteria : Correlation allelic expression level-phenotype Method : In Marfan patients with a FBN1 nul allele, FBN1 RNA will be extracted from a fibroblast culture. Allelic FBN1 expression level will be performed by quantitative RT-PCR and then compared with clinical evaluation.

Number of subjects : 160 subjects, 45 Marfan patients in 15 independent families, 5 patients with the same mutation, 30 with a private mutation leading to a nul allele and 80 non Marfan subjects.

Perspectives : To search the predictive factors of severity in order to ameliorate precocity of taking care.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman > 18 years old
* With a mutation in FBN1 gene
* Has signed an informed consent form

Exclusion Criteria:

-No affiliated to a Healthcare System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
FBN1 expression level | 6 months
  Evaluation in Marfan patients, of FBN1 expression level (non-mutated or mutated allele) compared to the clinical expression of the disease in idividuals

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Stheneur, PHD, MD, Principal Investigator — Hôpital Bichat, AP-HP
Locations (1):
- Centre de Reference Maladie de Marfan Et Apparente, Paris, Île-de-France Region, France